CLINICAL TRIAL: NCT03794804
Title: Double-blind, Randomized, Parallel-group, Placebo-controlled Study to Evaluate Efficacy of CMS008618 for Common Cold
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Enzymatica AB (Industry)
Collaborators: Analyze & Realize (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 008618
Record Dates: First submitted 2019-01-03; First posted 2019-01-07 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Common Cold
MeSH Terms: conditions — Common Cold

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ColdZyme (Active Comparator): ColdZyme® Mouth Spray. The IP should be applied every second hour up to 6 times, with each time 2 sprays (1 dose) per occasion.
  The IP use should start when following conditions have been fulfilled:
  * Answering "Yes" to either of the questions in the subject daily diary: "Do you think/feel you have a cold?" or "Do you think/feel you are coming down with a cold (might be having the first signs of cold)?" AND
  * A Jackson score of at least 1 in the subject's cold diary (mild = present, but not disturbing or irritating) for any symptom except headache
  The IP should be used until 2 days after the subject is symptom free (=answering "No" to the question "Do you think that you are still sick with this respiratory infection?" for 2 days in a row), but not longer than 10 days in total.
  Interventions: Device: ColdZyme
- Placebo (Placebo Comparator): Water based mouth spray manufactured to be similar to ColdZyme® Mouth Spray. The IP should be applied every second hour up to 6 times, with each time 2 sprays (1 dose) per occasion.
  The IP use should start when following conditions have been fulfilled:
  * Answering "Yes" to either of the questions in the subject daily diary: "Do you think/feel you have a cold?" or "Do you think/feel you are coming down with a cold (might be having the first signs of cold)?" AND
  * A Jackson score of at least 1 in the subject's cold diary (mild = present, but not disturbing or irritating) for any symptom except headache
  The IP should be used until 2 days after the subject is symptom free (=answering "No" to the question "Do you think that you are still sick with this respiratory infection?" for 2 days in a row), but not longer than 10 days in total.
  Interventions: Device: ColdZyme Placebo

INTERVENTIONS:
Device: ColdZyme — ColdZyme® Mouth Spray, a CE -marked device with the following composition of the spray solution: glycerol, purified water, cod trypsin, ethanol (<1 %), calcium chloride, trometamol and menthol.
  ColdZyme is a non-sterile mouth spray packaged in a primary container consisting of a 20 ml semi-transparent plastic bottle, pump, actuator (spray nozzle) and an actuator terminal cap.
  Arms: ColdZyme
Device: ColdZyme Placebo — The placebo mouth spray solution has the following composition: ethanol (<1 %), menthol and water. The placebo mouth spray is packaged in a primary container consisting of a 20 ml semitransparent plastic bottle, pump, actuator (spray nozzle) and an actuator terminal cap.
  Arms: Placebo

SUMMARY:
This study evaluates the impact of ColdZyme® Mouth Spray on quality of life during common cold. Half of the participants will receive ColdZyme® Mouth Spray, half will receive a placebo device.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women
2. Age 18 to 70 years old
3. Increased risk for common cold (at least 3 self-reported occurences of common cold within the last 12 months prior to V1) but generally in good health
4. Readiness to comply with trial procedures, including in particular:

   * Use of IP as recommended
   * Filling in diary
   * Keeping habitual life-style, including diet and physical activity level
   * No use of products that may influence the study outcome (e.g. immune suppressants/immune stimulants including natural health products, analgesics/anti-rheumatics, anti-phlogistics, anti-tussives/expectorants, mouth or throat therapeutics, decongestants, antibiotics, anti-histaminergic drugs, nasal drops/spray) during the study (except for the defined "rescue" treatment)
5. Women of child-bearing potential:

   * Have to agree to use appropriate contraception methods
   * Negative pregnancy testing (beta human chorionic gonadotropin test in urine) at V1

Participation is based upon written informed consent by the participant following written and oral information by the investigator regarding nature,

Exclusion Criteria:

1. Known allergy or hypersensitivity to the components of the investigational product
2. History and/or presence of clinically significant condition/ disorder (self-reported), which per investigator's judgement could interfere with the results of the study or the safety of the subject, e.g.:

   * Nasal disorder (e.g. polyposis, relevant septal deviation, ulcer etc.) and/or reconstructive surgery
   * Asthma, chronic obstructive lung disease or any other acute/chronic airways disease/disorder (e.g. chronic cough of any origin)
   * Acute psychiatric disorders
   * Any other acute/chronic serious organ or systemic diseases
3. Influenza vaccination within the last 3 months prior to V1 and during the study
4. Regular use of products that may influence the study outcome (e.g. immune suppressants/immune stimulants including natural health products, analgesics/anti-rheumatics, anti-phlogistics, antitussives/ expectorants, mouth or throat therapeutics, decongestants, antibiotics, anti-histaminergic drugs, nasal drops/spray) within the last 4 weeks prior to V1
5. Pregnancy or nursing
6. History of (in the past 12 months prior to V1) or current abuse of drugs, alcohol or medication
7. Participation in the present study of a person living in the same household as the subject
8. Inability to comply with study requirements according to investigator's judgement
9. Participation in another clinical study in the 30 days prior to V1 and during the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 701 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2019-06-26 (Actual)

PRIMARY OUTCOMES:
WURSS-21 QoL sub score | Days 1-8 (day 1 is the first day of symptoms)
  The primary endpoint is the AUC of Wisconsin Upper Respiratory Symptom Survey (WURSS-21) Quality of Life composite subscore during first 8 days of symptoms, to be assessed in comparison between verum and placebo.

SECONDARY OUTCOMES:
1. Composite daily severity of all symptoms within the Jackson score | Days 1-8 (day 1 is the first day of symptoms)
  The first major secondary endpoint: AUC days 1-8 composite daily severity of all symptoms within the Jackson score (mean of morning and evening) (day 1 is the first day of symptom recording)
2. Exposure to any concomitant treatment (including natural health products) that may affect common cold symptoms | Days 1-4 (day 1 is the first day of symptoms)
  The second major secondary endpoint: Exposure to any concomitant treatment (including natural health products) that may affect common cold symptoms - immune suppressants/immune stimulants, analgesics/ anti-rheumatics, anti-phlogistics, antitussives/ expectorants, mouth or throat therapeutics, decongestants, antibiotics, anti-histaminergic drugs, nasal drops/spray or any medication/treatment known to affect common cold symptoms - at any dose, expressed as number of days with concomitant treatment during the first 4 days for each subject (based on diary data).
Other secondary endpoints: AUC days 1-8 for each single WURSS-21 QoL subscore item | Days 1-8 (day 1 is the first day of symptoms)
  AUC days 1-8 for each single WURSS-21 QoL subscore item
AUC days 1-8 composite daily severity of all local symptoms within the Jackson score (mean of morning and evening) | Days 1-8 (day 1 is the first day of symptoms)
  AUC days 1-8 composite daily severity of all local symptoms within the Jackson score (mean of morning and evening) item
AUC days 1-8 composite daily severity of each individual symptom of the Jackson score (mean of morning and evening) | Days 1-8 (day 1 is the first day of symptoms)
  AUC days 1-8 composite daily severity of all local symptoms within the Jackson score (mean of morning and evening) item
Frequency of subjects with use of concomitant treatment that may affect common cold symptoms or any medication/treatment known to affect common cold symptoms - at any dose | Days 1-4
  Frequency of subjects with use of concomitant treatment (including natural health products) that may affect common cold symptoms - immune suppressants/immune stimulants, analgesics/anti-rheumatics, anti-phlogistics, antitussives/expectorants, mouth or throat therapeutics, decongestants, antibiotics, anti-histaminergic drugs, nasal drops/spray or any medication/treatment known to affect common cold symptoms - at any dose
Assessment of duration of first intense phase | From enrolment through study completion, maximum 16 weeks
  Assessment of duration of first intense phase, expressed as number of days from start of treatment until scoring <5 in total Jackson score
Assessment of symptom intensity | Days 1-4
  Assessment of symptom intensity, expressed as mean total Jackson score days 1-4
Assessment of symptom sore throat per Sore Throat Scale | Days 1-8
  Assessment of symptom sore throat per Sore Throat Scale, expressed as AUC days 1-8
Percentage of subjects with confirmed common cold at Visit 2 | 1-3 days after symptom start
  Percentage of subjects with confirmed common cold at Visit 2 (from all subjects with V2), which should take place within 1-3 days after symptom start
Global evaluation of efficacy by subjects and investigators at study end | From enrolment through study completion, maximum 16 weeks
  Global evaluation of efficacy by subjects and investigators at study end, 4-point categorical scale: "very good", "good", "moderate" and "poor"

OTHER OUTCOMES:
Safety endpoint: Physical examination | From enrolment through study completion, maximum 16 weeks
  Physical examination: standard clinical examination of the gastrointestinal tract, cardiovascular system, eyes, respiratory tract, lymph nodes, musculoskeletal system, neurological functions, urogenital tract, thyroid gland and skin.
Safety endpoint: Vital signs | From enrolment through study completion, maximum 16 weeks
  Vital signs: blood pressure (mmHg)
Safety endpoint: Vital signs | From enrolment through study completion, maximum 16 weeks
  Vital signs: pulse rate (bpm)
Safety endpoint: Global evaluation of tolerability by subjects and investigators | From enrolment through study completion, maximum 16 weeks
  Global evaluation of tolerability by subjects and investigators at study end, 4-point categorical scale: "very good", "good", "moderate" and "poor"
Safety endpoint: Assessment of adverse events | From enrolment through study completion, maximum 16 weeks
  Assessment of adverse events throughout the study
Safety endpoint: Assessment of device deficiencies | From enrolment through study completion, maximum 16 weeks
  Assessment of device deficiencies at V2 and V3

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Uebelhack, Prof. Dr. med., Principal Investigator — analyze & realize GmbH
Locations (10):
- Germany (10):
  - analyze & realize GmbH, Berlin
  - emovis GmbH, Berlin
  - Klinische Forschung Berlin-Mitte GmbH, Berlin
  - Klinische Forschung Berlin, Berlin
  - Polikum Institut GmbH, Berlin
  - Praxis Frau Barbara Grube, Berlin
  - Thomas Wünsche, Berlin
  - BioTeSys GmbH, Esslingen am Neckar
  - Praxis Dr. med. Gudrun Ruhland, Koßdorf
  - SIBAmed Studienzentrum GmbH und Co. KG, Leipzig

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported, after deidentification (text, tables, figures, and appendices) will be shared with researchers who provide a methodologically sound proposal, to achieve aims in the approved proposal.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Individual participant data that underlie the results reported, after deidentification (text, tables, figures, and appendices) will be shared with researchers who provide a methodologically sound proposal, to achieve aims in the approved proposal. Proposals should be directed to fredrik.lindberg@enzymatica.com. To gain access, data requestors will need to sign a data access agreement.